CLINICAL TRIAL: NCT00892489
Title: Pivotal Bioequivalence Study With 15 mg ER OROS Paliperidone Comparing the Phase 3 Formulation With the To-be-marketed Formulation and Evaluation of Food Effect on the to be Marketed Formulation in Healthy Male Subjects
Brief Title: A Bioequivalence Study of 15 mg ER OROS Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR004213
Record Dates: First submitted 2008-12-18; First posted 2009-05-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, Mood disorders, Antipsychotics; ER OROS Paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: ER OROS Paliperidone

SUMMARY:
The purpose of this study is to evaluate the bioequivalence between the Phase 3 and the to-be-marketed formulations of extended release (ER) OROS paliperidone and to evaluate the effect of food on the highest to be marketed tablet strength. Additionally, the safety and tolerability of the treatments in healthy volunteers will be assessed.

DETAILED DESCRIPTION:
This study is designed as a single-center, open-label, randomized, 3 treatment-period, crossover study in healthy male adults. The study consists of a screening phase and an open-label treatment phase during which each volunteer will receive 3 treatments of study drug in a random order and separated by a washout period of 10 to 14 days. Treatment A consists of a single oral dose of 15 mg ER OROS paliperidone Phase 3 formulation in the fasted state; Treatment B consists of a single oral dose of 15 mg ER OROS paliperidone to-be-marketed formulation in fasted state; and Treatment C consists of a single oral dose of 15 mg ER OROS paliperidone to-be-marketed formulation after consumption of a high-fat breakfast. There are slight formulation differences between the ER OROS paliperidone formulation that was used in Phase 3 efficacy studies and the formulation that is intended to be marketed. What is more important, however, is that the highest tablet strength used in Phase 3 and the tablet strength that is planned for the market as commercial formulation are different. For Phase 3 studies, 9 mg was the highest tablet strength and the highest dose of 15 mg was administered as 2 tablets of 3 mg and 1 tablet of 9 mg. The highest to-be-marketed tablet strength is 15 mg. This study is designed to demonstrate the bioequivalence between the Phase 3 formulation and the highest tablet strength of the to-be-marketed formulation and to assess the effect of food on the highest to-be-marketed tablet strength. Safety and tolerability will be monitored throughout the study. All volunteers will receive each of the following 3 treatments in the order specified by the random assignment:Treatment A, oral ER OROS paliperidone Phase 3 formulation as 2 tablets of 3 mg and 1 tablet of 9 mg in the fasted state; Treatment B, oral ER OROS paliperidone to-be-marketed formulation as 1 tablet of 15 mg in the fasted state; Treatment C, oral ER OROS paliperidone to-be-marketed formulation as 1 tablet of 15 mg after a high-fat breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (weight [kg]/height [m²]) of 18 to 28 kg/m², inclusive
* Have a supine (after 5 minutes rest) blood pressure between the range of 100 to 140 mmHg systolic, inclusive, and 50 to 90 mmHg diastolic, inclusive
* Healthy on the basis of a prestudy physical examination, medical history, ECG, and the laboratory results of serum chemistry, hematology and urinalysis performed within 21 days before the first dose. If the results of the serum chemistry, hematology or urinalysis testing are not within the laboratory's reference ranges the volunteer can be included only if the investigator judges that the deviations are not clinically significant. For renal function tests, the values must be within the normal laboratory reference ranges.

Exclusion Criteria:

* Drug allergy to risperidone, paliperidone, or any of its excipients
* Known allergy or history of significant hypersensitivity to heparin, in case a heparin lock will be used
* Recent history of alcohol or substance abuse, a positive test result for the urine drug screen at screening or upon admittance to the testing facility or a positive result for the alcohol urine test upon admittance to the testing facility
* Relevant history or presence of any cardiovascular (including myocardial infarct or cardiac arrhythmia), respiratory, neurologic (including seizures), psychiatric, renal, hepatic, gastrointestinal (including surgeries, severe gastrointestinal narrowing, and malabsorption problems), endocrine, hematologic or immunologic disease
* History of any cancer, with the exception of basal cell carcinoma
* At screening, has a sustained decrease of >20 mmHg in systolic blood pressure or a decrease of >10 mmHg in diastolic blood pressure after standing for at least 2 minutes that is not associated with an increase of >15 beats per minute (bpm) in heart rate
* Bradycardia (heart rate <50 bpm) as determined by screening ECG
* History of or a positive test result for any of the serology tests (hepatitis B, C, and HIV)
* History of smoking or use of nicotine-containing substances within the last 2 months, as determined by medical history and/or volunteer's verbal report. Volunteers must agree to refrain from use throughout the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2004-07; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the bioequivalence between the Phase 3 and the to-be-marketed formulations of ER OROS paliperidone and to evaluate the effect of food on the highest to-be-marketed tablet strength

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the treatments in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A bioequivalence study of 15 mg ER OROS paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=568&filename=CR004213_CSR.pdf